CLINICAL TRIAL: NCT03352986
Title: A Substudy of the CADRE Study: Determination of Clinical Markers in Patients With Extreme Sickle Cell Disease Phenotype
Brief Title: Substudy of CADRE: for People With Extreme Phenotype: BIOCADRE
Acronym: BIOCADRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiologie et Développement (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 003
Record Dates: First submitted 2017-10-10; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; anemia; Africa
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3 ml of saliva for DNA extraction (sample with DNA) and 2 ml of plasma (sample with no DNA) are taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- osteonecrosis: Sickle cell patients with osteonecrosis as a vascular main complication
  Interventions: Biological: biological analysis; Other: peripheral arterial tonometry
- leg ulcer: Sickle cell patients with leg ulcer as a vascular main complication
  Interventions: Biological: biological analysis; Other: peripheral arterial tonometry
- microalbuminuria: Sickle cell patients with microalbuminuria as a vascular main complication
  Interventions: Biological: biological analysis; Other: peripheral arterial tonometry
- pulmonary hypertension: Sickle cell patients with pulmonary hypertension as a vascular main complication
  Interventions: Biological: biological analysis; Other: peripheral arterial tonometry
- stroke: Sickle cell patients with strocke as a vascular main complication
  Interventions: Biological: biological analysis; Other: peripheral arterial tonometry
- priapism: Sickle cell patients with priapism as a vascular main complication
  Interventions: Biological: biological analysis; Other: peripheral arterial tonometry

INTERVENTIONS:
Biological: biological analysis — biological analysis will be performed in the 6 groups of patients
Other: peripheral arterial tonometry — peripheral arterial tonometry will be performed in the 6 groups of patients

SUMMARY:
BIOCADRE is a CADRE substudy and aims to characterize more precisely the sickle cell patients with extreme phenotype.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is the most frequent monogenic disease in the world, due to a unique mutation on the β-globin gene. Most affected individuals live in sub-Saharan Africa, yet, the natural history of the disease in Africa remains largely unknown. SCD usually presents in childhood and is characterized by the association of a chronic hemolytic anemia with episodes of acute vaso-occlusive events and progressive vascular organ damage. SCD is now widely recognized as a vascular disease with marked endothelial dysfunction. Hemolysis probably plays a key role by reducing NO bioavailability, but other involved mechanisms are not fully understood.

The project aims at better understanding SCD chronic vascular complications and in particular to explore extensively the different mechanisms associated with hemolysis. This will be addressed through both an epidemiological approach and a hypotheses-driven pathophysiological approach. On the one hand, a descriptive and analytic epidemiological study will isolate clusters of clinical, functional and usual biological phenotypes in SCD patients and look for new mechanistic and biological markers predictive of chronic vascular complications in SCD with SS phenotype. Investigators will specifically investigate i) microcirculation functions using peripheral arterial tonometry, ii) blood and plasma viscosities, iii) level of plasma blood cell derived microparticles, free hemoglobin, and the free heme content of erythrocytes-derived microparticles and expression of Duffy erythrocyte antigen, the unique erythroid receptor for chemokines. One the other hand, investigators will test novel markers and modifiers of hemolysis and heme metabolism and assess their relationship with inflammation and vascular phenotypes.These different biomarkers will be compared between the selected subgroups of patients with extreme vascular phenotype.

Methods: The project involves a transversal case control study, nested in the CADRE cohort, recently built up by Partner 1 and African collaborators. CADRE is the largest ongoing epidemiological cohort, including 4,300 SCD patients and 1,000 controls in five west and central African countries, in which various chronic complications of SCD have already been registered. The present second phase study will be conducted in the centres of Dakar and Bamako. Patients' selection will be performed in the existing database to obtain 6 subgroups of 40 SS patients with one of the main vascular chronic complications or none of them, for a total of 240 patients. Selected patients will be recalled during one year in parallel in the 2 recruiting centres. Clinical phenotyping, usual biology, functional microvascular functions (peripheral arterial tonometry), and blood/plasma viscosities analyses will be performed in the African recruiting centres after training of technicians, PhD and MD students by the French partners. Plasma samples, microparticles and extracellular DNA, will be prepared and frozen for further analyses in the partner's laboratories. DNA will be collected for each subject. A principal component analysis will isolate clusters of clinical complications, functional and biological markers and a multivariate logistic regression will quantify the effect of these markers on the risk of vasculopathy, with adjustment on all known SCD modifying factors.

Expected results: 1) The identification of high risk SCD patients for chronic vascular complications using new biomarkers, 2) A better understanding of chronic vascular disease process at the mechanistic and biological (viscosity, hemolysis, erythrocyte derived microparticles, inflammatory cytokines and receptors) levels, 3) The identification of endophenotypes and constitution of DNA bank for further genetic studies.

ELIGIBILITY:
Inclusion Criteria:

* sickle cell patients with extreme phenotypes: SS-hemoglobin

Exclusion Criteria:

* transfusion in the previous 2 months
* vaso-occlusive crisis in the previous 15 days
* infection in the previous 8 days

Min Age: 10 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population is sickle cell patients with extreme phenotypes (SS-hemoglobin) with a steady state.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Description of microcirculation by peripheral arterial tonometry | 1 year
  EndoPAT2000®, Itamar Medical Ltd,

SECONDARY OUTCOMES:
Measure of blood viscosities | 1 year
  In whole blood by viscosimeter
Dosage of microparticles | 1 year
  In plasma: microparticles of erythrocytic, platelet, monocytic, neutrophilic and endothelial origin by flow cytometry
Determination of free hemoglobin | 1 year
  In plasma
Measurement of neutrophil extracellular trap (NET) | 1 year
  In plasma
Measurement of proinflammatory cytokines by ELISA | 1 year
  In plasma by ELISA
Genotyping of the alpha-globin gene associated with persistence of fetal hemoglobin | 1 year
  In saliva DNA
Genotyping of the polymorphisms associated with persistence of fetal hemoglobin | 1 year
  In saliva DNA

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Ranque, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (2):
- Centre de Recherches er de Lutte contre la Drépanocytose, Bamako, Mali
- Centre National de Transfusion Sanguine, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranque B, Menet A, Diop IB, Thiam MM, Diallo D, Diop S, Diagne I, Sanogo I, Kingue S, Chelo D, Wamba G, Diarra M, Anzouan JB, N'Guetta R, Diakite CO, Traore Y, Legueun G, Deme-Ly I, Belinga S, Boidy K, Kamara I, Tharaux PL, Jouven X. Early renal damage in patients with sickle cell disease in sub-Saharan Africa: a multinational, prospective, cross-sectional study. Lancet Haematol. 2014 Nov;1(2):e64-73. doi: 10.1016/S2352-3026(14)00007-6. Epub 2014 Oct 28. PMID 27030156
- [Background] Ranque B, Menet A, Boutouyrie P, Diop IB, Kingue S, Diarra M, N'Guetta R, Diallo D, Diop S, Diagne I, Sanogo I, Tolo A, Chelo D, Wamba G, Gonzalez JP, Abough'elie C, Diakite CO, Traore Y, Legueun G, Deme-Ly I, Faye BF, Seck M, Kouakou B, Kamara I, Le Jeune S, Jouven X. Arterial Stiffness Impairment in Sickle Cell Disease Associated With Chronic Vascular Complications: The Multinational African CADRE Study. Circulation. 2016 Sep 27;134(13):923-33. doi: 10.1161/CIRCULATIONAHA.115.021015. Epub 2016 Aug 31. PMID 27582423
- [Background] Kato GJ, Gladwin MT, Steinberg MH. Deconstructing sickle cell disease: reappraisal of the role of hemolysis in the development of clinical subphenotypes. Blood Rev. 2007 Jan;21(1):37-47. doi: 10.1016/j.blre.2006.07.001. Epub 2006 Nov 7. PMID 17084951
- [Background] Hebbel RP. Reconstructing sickle cell disease: a data-based analysis of the "hyperhemolysis paradigm" for pulmonary hypertension from the perspective of evidence-based medicine. Am J Hematol. 2011 Feb;86(2):123-54. doi: 10.1002/ajh.21952. PMID 21264896
- [Background] Tharaux PL. Endothelin in renal injury due to sickle cell disease. Contrib Nephrol. 2011;172:185-199. doi: 10.1159/000328699. Epub 2011 Aug 30. PMID 21893999
- [Background] Connes P, Lamarre Y, Hardy-Dessources MD, Lemonne N, Waltz X, Mougenel D, Mukisi-Mukaza M, Lalanne-Mistrih ML, Tarer V, Tressieres B, Etienne-Julan M, Romana M. Decreased hematocrit-to-viscosity ratio and increased lactate dehydrogenase level in patients with sickle cell anemia and recurrent leg ulcers. PLoS One. 2013 Nov 4;8(11):e79680. doi: 10.1371/journal.pone.0079680. eCollection 2013. PMID 24223994
- [Background] Bunn HF, Nathan DG, Dover GJ, Hebbel RP, Platt OS, Rosse WF, Ware RE. Pulmonary hypertension and nitric oxide depletion in sickle cell disease. Blood. 2010 Aug 5;116(5):687-92. doi: 10.1182/blood-2010-02-268193. Epub 2010 Apr 15. PMID 20395414
- [Background] Kato GJ, McGowan V, Machado RF, Little JA, Taylor J 6th, Morris CR, Nichols JS, Wang X, Poljakovic M, Morris SM Jr, Gladwin MT. Lactate dehydrogenase as a biomarker of hemolysis-associated nitric oxide resistance, priapism, leg ulceration, pulmonary hypertension, and death in patients with sickle cell disease. Blood. 2006 Mar 15;107(6):2279-85. doi: 10.1182/blood-2005-06-2373. Epub 2005 Nov 15. PMID 16291595
- [Background] Kato GJ, Hebbel RP, Steinberg MH, Gladwin MT. Vasculopathy in sickle cell disease: Biology, pathophysiology, genetics, translational medicine, and new research directions. Am J Hematol. 2009 Sep;84(9):618-25. doi: 10.1002/ajh.21475. PMID 19610078
- [Background] Nouraie M, Lee JS, Zhang Y, Kanias T, Zhao X, Xiong Z, Oriss TB, Zeng Q, Kato GJ, Gibbs JS, Hildesheim ME, Sachdev V, Barst RJ, Machado RF, Hassell KL, Little JA, Schraufnagel DE, Krishnamurti L, Novelli E, Girgis RE, Morris CR, Rosenzweig EB, Badesch DB, Lanzkron S, Castro OL, Goldsmith JC, Gordeuk VR, Gladwin MT; Walk-PHASST Investigators and Patients. The relationship between the severity of hemolysis, clinical manifestations and risk of death in 415 patients with sickle cell anemia in the US and Europe. Haematologica. 2013 Mar;98(3):464-72. doi: 10.3324/haematol.2012.068965. Epub 2012 Sep 14. PMID 22983573
- [Background] Aessopos A, Farmakis D, Tsironi M, Diamanti-Kandarakis E, Matzourani M, Fragodimiri C, Hatziliami A, Karagiorga M. Endothelial function and arterial stiffness in sickle-thalassemia patients. Atherosclerosis. 2007 Apr;191(2):427-32. doi: 10.1016/j.atherosclerosis.2006.04.015. Epub 2006 May 18. PMID 16712855
- [Background] Tharaux PL, Girot R, Kanfer A, Dussaule JC, Gaitz JP, Tribout L, Baudot N, Vayssairat M. Cutaneous microvascular blood flow and reactivity in patients with homozygous sickle cell anaemia. Eur J Haematol. 2002 Jun;68(6):327-31. doi: 10.1034/j.1600-0609.2002.02701.x. PMID 12225389
- [Background] van Beers EJ, Schaap MC, Berckmans RJ, Nieuwland R, Sturk A, van Doormaal FF, Meijers JC, Biemond BJ; CURAMA study group. Circulating erythrocyte-derived microparticles are associated with coagulation activation in sickle cell disease. Haematologica. 2009 Nov;94(11):1513-9. doi: 10.3324/haematol.2009.008938. Epub 2009 Oct 8. PMID 19815831
- [Background] Donadee C, Raat NJ, Kanias T, Tejero J, Lee JS, Kelley EE, Zhao X, Liu C, Reynolds H, Azarov I, Frizzell S, Meyer EM, Donnenberg AD, Qu L, Triulzi D, Kim-Shapiro DB, Gladwin MT. Nitric oxide scavenging by red blood cell microparticles and cell-free hemoglobin as a mechanism for the red cell storage lesion. Circulation. 2011 Jul 26;124(4):465-76. doi: 10.1161/CIRCULATIONAHA.110.008698. Epub 2011 Jul 11. PMID 21747051
- [Background] Nebor D, Bowers A, Connes P, Hardy-Dessources MD, Knight-Madden J, Cumming V, Reid M, Romana M. Plasma concentration of platelet-derived microparticles is related to painful vaso-occlusive phenotype severity in sickle cell anemia. PLoS One. 2014 Jan 24;9(1):e87243. doi: 10.1371/journal.pone.0087243. eCollection 2014. PMID 24475257
- [Background] Camus SM, Gausseres B, Bonnin P, Loufrani L, Grimaud L, Charue D, De Moraes JA, Renard JM, Tedgui A, Boulanger CM, Tharaux PL, Blanc-Brude OP. Erythrocyte microparticles can induce kidney vaso-occlusions in a murine model of sickle cell disease. Blood. 2012 Dec 13;120(25):5050-8. doi: 10.1182/blood-2012-02-413138. Epub 2012 Sep 13. PMID 22976952
- [Background] Reiter CD, Wang X, Tanus-Santos JE, Hogg N, Cannon RO 3rd, Schechter AN, Gladwin MT. Cell-free hemoglobin limits nitric oxide bioavailability in sickle-cell disease. Nat Med. 2002 Dec;8(12):1383-9. doi: 10.1038/nm1202-799. Epub 2002 Nov 11. PMID 12426562
- [Background] Turhan A, Weiss LA, Mohandas N, Coller BS, Frenette PS. Primary role for adherent leukocytes in sickle cell vascular occlusion: a new paradigm. Proc Natl Acad Sci U S A. 2002 Mar 5;99(5):3047-51. doi: 10.1073/pnas.052522799. PMID 11880644
- [Background] Chaar V, Picot J, Renaud O, Bartolucci P, Nzouakou R, Bachir D, Galacteros F, Colin Y, Le Van Kim C, El Nemer W. Aggregation of mononuclear and red blood cells through an alpha4beta1-Lu/basal cell adhesion molecule interaction in sickle cell disease. Haematologica. 2010 Nov;95(11):1841-8. doi: 10.3324/haematol.2010.026294. Epub 2010 Jun 18. PMID 20562314
- [Background] El Nemer W, Wautier MP, Rahuel C, Gane P, Hermand P, Galacteros F, Wautier JL, Cartron JP, Colin Y, Le Van Kim C. Endothelial Lu/BCAM glycoproteins are novel ligands for red blood cell alpha4beta1 integrin: role in adhesion of sickle red blood cells to endothelial cells. Blood. 2007 Apr 15;109(8):3544-51. doi: 10.1182/blood-2006-07-035139. Epub 2006 Dec 7. PMID 17158232
- [Background] Chen G, Zhang D, Fuchs TA, Manwani D, Wagner DD, Frenette PS. Heme-induced neutrophil extracellular traps contribute to the pathogenesis of sickle cell disease. Blood. 2014 Jun 12;123(24):3818-27. doi: 10.1182/blood-2013-10-529982. Epub 2014 Mar 11. PMID 24620350
- [Background] Tournamille C, Colin Y, Cartron JP, Le Van Kim C. Disruption of a GATA motif in the Duffy gene promoter abolishes erythroid gene expression in Duffy-negative individuals. Nat Genet. 1995 Jun;10(2):224-8. doi: 10.1038/ng0695-224. PMID 7663520
- [Background] Connes P, Lamarre Y, Waltz X, Ballas SK, Lemonne N, Etienne-Julan M, Hue O, Hardy-Dessources MD, Romana M. Haemolysis and abnormal haemorheology in sickle cell anaemia. Br J Haematol. 2014 May;165(4):564-72. doi: 10.1111/bjh.12786. Epub 2014 Feb 24. PMID 24611951
- [Background] Bollee G, Flamant M, Schordan S, Fligny C, Rumpel E, Milon M, Schordan E, Sabaa N, Vandermeersch S, Galaup A, Rodenas A, Casal I, Sunnarborg SW, Salant DJ, Kopp JB, Threadgill DW, Quaggin SE, Dussaule JC, Germain S, Mesnard L, Endlich K, Boucheix C, Belenfant X, Callard P, Endlich N, Tharaux PL. Epidermal growth factor receptor promotes glomerular injury and renal failure in rapidly progressive crescentic glomerulonephritis. Nat Med. 2011 Sep 25;17(10):1242-50. doi: 10.1038/nm.2491. PMID 21946538
- [Background] Sabaa N, de Franceschi L, Bonnin P, Castier Y, Malpeli G, Debbabi H, Galaup A, Maier-Redelsperger M, Vandermeersch S, Scarpa A, Janin A, Levy B, Girot R, Beuzard Y, Leboeuf C, Henri A, Germain S, Dussaule JC, Tharaux PL. Endothelin receptor antagonism prevents hypoxia-induced mortality and morbidity in a mouse model of sickle-cell disease. J Clin Invest. 2008 May;118(5):1924-33. doi: 10.1172/JCI33308. PMID 18382768